CLINICAL TRIAL: NCT04450498
Title: A Phase IV Randomized, Observer-blind, Controlled Study to Demonstrate Non-inferior Immunogenicity of Yuxi Walvax MPV ACYW® Vaccine as Compared to Sanofi Pasteur Menactra® Vaccine in Healthy Subjects Aged 2-10 Years
Brief Title: A Study to Demonstrate Non-inferior Immunogenicity of Yuxi Walvax MPV ACYW® Vaccine in Healthy Subjects Aged 2-10 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MPV ACYW-004
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Neisseria Meningitides Meningitis
Keywords: Neisseria Meningitidis; Non-inferior immunogenicity; Safety
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Intervention Model Description: At Day 0, eligible subjects will be randomized in a 1:1 ratio into either Walvax MPV ACYW® vaccine group (130 subjects) or Sanofi Pasteur Menactra ® vaccine group (130 subjects). A randomization list containing subject numbers and vaccine group assignments will be provided to the investigator. Each participant will receive a single intramuscular injection of one of the two vaccines either MPV ACYW® vaccine or Menactra ® vaccine according to the vaccine group assignment and will be followed up for one month for immunogenicity evaluation and for 6 months for safety evaluation.
Who Masked: Investigator
Masking Description: The study will be carried out in an observer blind fashion until database is locked with data collected until Day 30 (Visit 3) after vaccination. The clinical study material, i.e. vaccine packs, will be packaged and encoded according to the randomization list (see Appendix B for example of vaccine labels). At study site, the investigator will assign unblinded designated person(s) responsible for vaccine handling, administration ("Vaccinator") and accountability to ensure that blinding is protected throughout the study procedures and that no other site personnel involved in the conduct of the study has access to the information. After assessment of eligibility of a new subject, the investigator will complete a form that the subject will take to the "vaccinator". The "vaccinator" will administer the vaccine according to the randomization list to the subject without informing neither the subject nor the investigator of the randomization group, i.e. the nature of the vaccine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walvax MPV ACYW® vaccine group (Experimental)
  Interventions: Biological: Yuxi Walvax MPV ACYW® vaccine
- Sanofi Pasteur Menactra® vaccine group (Active Comparator)
  Interventions: Biological: Sanofi Pasteur Menactra® vaccine

INTERVENTIONS:
Biological: Yuxi Walvax MPV ACYW® vaccine — Walvax MPV ACYW vaccine is a sterile formulation of polysaccharide A,C,Y,W-135. One dose of 0.5 mL contains 50 µg of each A,C,Y,W-135 purified polysaccharide. The vaccine is presented in two vials: one containing the lyophilized cake of A,C,Y,W purified polysaccharides and the other the sterile water for injection as diluent. After reconstitution the one dose of 0.5 mL is ready for subcutaneous injection. The antigen content is similar to other internationally marketed polysaccharide vaccines that have been in use for decades as Menomune® Sanofi and Mencevax® Pfizer , all containing 50 µg of each A,C,Y,W purified polysaccharide that as one dose schedule are recommended for use in subjects > 2 years of age and have shown to be safe and immunogenic.
  Arms: Walvax MPV ACYW® vaccine group
Biological: Sanofi Pasteur Menactra® vaccine — The vaccine presentation is a full liquid formulation in a single dose of 0.5 mL with the following composition: Meningococcal group A polysaccharide 4 µg; Meningococcal group C polysaccharide 4 µg; Meningococcal group Y polysaccharide 4 µg; Meningococcal group W polysaccharide 4 µg; Diphtheria toxoid protein total 48 µg; Sodium phosphate 0.7 mg; Sodium chloride 4.35 mg.
  Arms: Sanofi Pasteur Menactra® vaccine group

SUMMARY:
This is a phase IV, single-center, observer-blind, randomized, controlled vaccine trial in 2 to 10 years old healthy subjects. Each participant will receive a single intramuscular injection of one of the two vaccines either MPV ACYW® vaccine or Menactra ® vaccine according to the vaccine group assignment and will be followed up for one month for immunogenicity evaluation and for 6 months for safety evaluation.

Statistical Hypothesis:

H0: Seroconversion rate of test group is inferior to that of control group HA: Seroconversion rate of test group is non-inferior to that of control group Sample size calculation: the sample size was calculated based on non-inferiority test with alpha level of 0.025 and 80% power, assuming seroconversion rate in control group was 95% with non-inferiority margin at 10%. The sample size required for the study is 124 per arm. After adjusting for 5% drop-out, the final sample size required is 130 per arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 10 years of age (both included)
* Written informed consent obtained from the mother, father, or guardian of the child.
* Free of obvious health problems and be fully vaccinated according local EPI schedule as established by medical history including physical examination and clinical judgment of the investigator.
* Mother, father, or guardian capable and willing to bring their child or to receive home visits for their child for all follow-up visits.
* Residence in the study area during the study period.

Exclusion Criteria:

* Vaccination against group A,C,Y,W Neisseria meningitidis in the previous 3 months
* History of allergic disease or known hypersensitivity to any component of the two study vaccines.
* History of serious adverse reactions following administration of vaccines included in the local program of immunization.
* Administration of any other vaccine within 30 days prior to administration of study vaccines or planned vaccination during the first four weeks after the study vaccination.
* Use of any investigational or nonregistered product within 60 days prior to the administration of study vaccines.
* Administration of immunoglobulins and/or any blood products or planned administration during the study participation period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying agents since birth (including systemic or inhaled corticosteroids, this means prednisone, or equivalent, ≥0.5 mg/kg/day; topical steroids are allowed).
* A family history of congenital or hereditary immunodeficiency.
* History of meningitis or seizures, or any neurological disorder, convulsions, or active tuberculosis.
* Major congenital defects or serious chronic illness, including malnutrition (i.e., weight less than or equal to 3 standard deviations below the mean for 2-5 years old) and immunodeficiency disorder (as per investigator's judgment)
* Acute disease at the time of enrollment (acute disease being defined as the presence of a moderate or severe illness with or without fever) resulting in a temporary exclusion.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history, physical examination, or laboratory tests, which in the opinion of the investigator might interfere with the well-being of the subject study objectives.
* Any condition or criterion that in the opinion of the investigator might compromise the well-being of the subject or the compliance with study procedures or interfere with the outcome of the study

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Antibody response at Day 30 post-vaccination | Day 30 post-vaccination
  Percentage of subjects with rSBA (Serum Bactericidal Activity using baby rabbit complement) titer ≥1:128 to A,C,Y,W meningococcal capsular polysaccharide in both vaccine groups 30 days after immunization

SECONDARY OUTCOMES:
Percentages of subjects with post-immunization local and systemic reactions within 7 days following vaccination in both vaccine groups | Day 7 post-vaccination
Percentages of subjects with reported Adverse Events within 30 days following vaccination in both vaccine groups | Day 30 post-vaccination
Percentages of subjects with reported SAEs within 6 months following vaccination in both vaccine groups | Day 30 to Day 180 post-vaccination (end of study visit)
rSBA Geometric mean antibody titers to A,C,Y,W meningococcal capsular polysaccharide in both vaccine groups | Day 30 post-vaccination
Percentage of subjects with rSBA titer ≥1:8 to A,C,Y,W meningococcal capsular polysaccharide in both vaccine groups 30 days after immunization | Day 30 post-vaccination
Seroconversion rates as defined by proportion of subjects with ≥ 4-fold increase 30 days after immunization with respect to baseline of rSBA antibodies to A,C,Y,W meningococcal capsular polysaccharide in both vaccine groups 30 days after immunization | Day 30 post-vaccination
Seroconversion rates as defined by proportion of subjects with ≥ 2-fold increase 30 days after immunization with respect to baseline of rSBA antibodies to A,C,Y,W meningococcal capsular polysaccharide in both vaccine groups | Day 30 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Samba O Sow, MD, MSc, Principal Investigator — Director General
Locations (1):
- Centre pour le Développement des Vaccins du Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sow SO, Tapia MD, Haidara FC, Diallo F, Traore Y, Traore A, Kodio M, Borrow R, Townsend-Payne K, Yuan L, Yang S, Shi L, Chen J, Fang G, Lin J, Hu R, Viviani S, Huang Z. Safety and immunogenicity of quadrivalent meningococcal polysaccharide vaccine (MPV ACYW135) compared with quadrivalent meningococcal conjugate vaccine (Menactra(R)) in Malian children. Hum Vaccin Immunother. 2023 Aug 1;19(2):2230829. doi: 10.1080/21645515.2023.2230829. Epub 2023 Jul 4. PMID 37401618